CLINICAL TRIAL: NCT02320929
Title: The Treatment of Purulent Flexor Tenosynovitis - is Postoperative Catheter Irrigation Necessary? a Prospective Randomized Trial.
Brief Title: The Treatment of Purulent Flexor Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Olli Leppänen, Researcher, M.D., Ph.D., Tampere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R14153
Record Dates: First submitted 2014-12-08; First posted 2014-12-19 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Tenosynovitis
Keywords: irrigation; tenosynovitis; purulent; closed-catheter; flexor tendon
MeSH Terms: conditions — Tenosynovitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraoperative irrigation only (Experimental): The infected tendon sheath is irrigated intraoperatively, the catheter is removed, and small rubber srains are left in small incisions.
  Interventions: Procedure: Intraoperative flexor tendon sheath irrigation
- Intra- and postoperative irrigation (Active Comparator): The infected tendon sheath is irrigated intraoperatively, the catheter is kept in place, the irrigation is continued postoperatively 3 times a day for 3 days.
  Interventions: Procedure: Intraoperative flexor tendon sheath irrigation; Procedure: Postoperative flexor tendon sheath irrigation

INTERVENTIONS:
Procedure: Intraoperative flexor tendon sheath irrigation
Procedure: Postoperative flexor tendon sheath irrigation
  Arms: Intra- and postoperative irrigation

SUMMARY:
This study evaluates the effect of postoperative intermittent closed-catheter irrigation on the recovery from the purulent flexor tenosynovitis. One group of patients suffering from acute purulent flexor tenosynovitis is treated using intraoperative irrigation only and the other group having both intra- and postoperative irrigation.

DETAILED DESCRIPTION:
The foundation of the successful management of purulent flexor tenosynovitis is the surgical debridement followed by an intravenous antibiotic treatment. Several surgical methods have been described to remove the purulent debris from the flexor tendon sheath. Closed-catheter irrigation involves irrigation of the tendon sheath from proximal to distal direction facilitated by two small incisions; one proximal to A1 pulley and one distal to A4 pulley. Lille et al. (J Hand Surg Br. 2000;25(3):304-307) conducted a retrospective study that implied that intraoperative closed-catheter irrigation without postoperative irrigation might be as effective as the combination of intra- and postoperative irrigation.

The hypothesis of this prospective randomized trial is that the intraoperative closed-catheter irrigation alone is as effective as the combination of intraoperative and postoperative intermittent closed-catheter irrigation in the treatment of purulent flexor tenosynovitis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of purulent flexor tenosynovitis with all four positive Kanavel's signs:

  * symmetric swelling of the entire digit
  * exquisite tenderness along the course of the tendon sheath
  * semiflexed posture of the digit
  * pain with attempted passive extension of the digit
* age over 18 years
* patient's willingness to participate in the study

Exclusion Criteria:

* High-pressure, foreign body or chemical injuries, which require open debridement
* prisoner, military serviceman, mental retardation or other factors which may affect one's decision making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Active range of movement of the most affected finger | 3 months postoperatively
  The total active range of movement is calculated as: (active flexion of MCPJ + PIPJ + DIPJ) - (extension deficit of MCPJ + PIPJ + DIPJ). MCPJ, metacarpophalangeal joint; PIPJ, proximal interphalangeal joint; DIPJ, distal interphalangeal joint.

SECONDARY OUTCOMES:
Need for reoperation | 3 months postoperatively

OTHER OUTCOMES:
QuickDASH score | 4 weeks and 3 months postoperatively
Pain at rest | 4 weeks and 3 months postoperatively
  Pain at rest (Visual analog scale)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Göransson, M.D., Ph.D., Study Chair — Chief surgeon, Department of Hand and Microsurgery, Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Leppanen OV, Jokihaara J, Kaivorinne A, Havulinna J, Goransson H. Protocol for an investigator-blinded, randomised, 3-month, parallel-group study to compare the efficacy of intraoperative tendon sheath irrigation only with both intraoperative and postoperative irrigation in the treatment of purulent flexor tenosynovitis. BMJ Open. 2015 Dec 15;5(12):e008824. doi: 10.1136/bmjopen-2015-008824. PMID 26671952